CLINICAL TRIAL: NCT05734144
Title: Two Institutes Experience In Laparo-Endoscopic Rendezvous Technique For Patients Undergoing Laparscopic Cholecystectomy For Stones In The Gallbladder And Bile Duct; A Prospective Randomized Comparative Clinical Trial
Brief Title: Two Institutes Experience in Laparo-Endoscopic Rendezvous Technique for Gallbladder and Bile Duct Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mohamed I Farid, assistant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 10129/20-11-2022
Record Dates: First submitted 2023-02-03; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Calculus; Gallbladder, With Cholecystitis
MeSH Terms: conditions — Calculi

STUDY DESIGN:
Intervention Model Description: This study was carried out on 432 patients with gall bladder stones and with suspected or confirmed CBDS at two centers 264 patients at the Gastrointestinal Surgery Unit in the Zagazig University Hospitals and 168 patients at gastroenterology surgery unite at ALAHRAR hospitals from January 2010 till May 2022. Patients were randomized divided into two equally groups, the first group was treated by a single-step procedure combining LC and IOES while the second (control) group was treated by 2-stage (sequential treatment) POES followed by LC.
Who Masked: Participant, Care Provider
Masking Description: both the participant patients and the surgeon had no knowledge about the chosen procedure and the choosen procedure were known by the investigator who told the surhgeon later which procedure to perform for the selected patient.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparo-endoscopic "rendezvous" technique (Active Comparator): the first group was treated by a single-step procedure combining LC and IOES
  Interventions: Procedure: The intraoperative ERCP has been performed immediately before LC
- POES followed by LC (Other): the second (control) group was treated by 2-stage (sequential treatment) POES followed by LC.
  Interventions: Procedure: POES followed by LC

INTERVENTIONS:
Procedure: The intraoperative ERCP has been performed immediately before LC — combination approach has been used to improve patient compliance and shorten hospital stays. The intraoperative ERCP has been performed immediately before Laparoscopic Cholecystectomy
  Arms: Laparo-endoscopic "rendezvous" technique
Procedure: POES followed by LC — Treatment in two stages, which combines a preoperative ES followed by LC (sequential treatment).
  Arms: POES followed by LC

SUMMARY:
The management of gallbladder stones (lithiasis) concomitant with bile duct stones is controversial. The management of CBD stones has evolved considerably since the advent of laparoscopic surgery. The more frequent approach is a two-stage procedure, with endoscopic sphincterotomy and stone removal from the bile duct followed by laparoscopic cholecystectomy. The laparoscopic-endoscopic rendezvous combines the two techniques in a single-stage operation. So the aim of this study was was to evaluate one-stage LC with intra-operative endoscopic sphincterotomy (IOES) vs two-stage pre-operative endoscopic sphincterotomy (POES) followed by LC for the treatment of cholecystocholedocholithiasis.

DETAILED DESCRIPTION:
This is two center study was carried out on 523 patients and completed in 436 patients with gall bladder stones and with suspected or confirmed CBDS at two gastroenterology center at zagazig first 264 patients at the Gastrointestinal Surgery Unit in the Zagazig University Hospitals and second 172 patients at gastroenterology unite at AL AHRAR hospital from January 2010 till April 2022. A single-step technique combining LC and IO-ERCP was used to treat them. To confirm the presence of CBDS, a laparoscopic intraoperative cholangiography (IOC) was performed. A soft-tipped guidewire was inserted into the duodenum through the cystic duct and papilla. Over the guide-wire, an endoscopic papillotomy was introduced. The stones were retrieved with a retrieval balloon after an IO-ERCP and endoscopic sphincterotomy. The length of the postoperative hospital stay, surgical operating time, surgical success rate, postoperative complications, and residual CBDS were all evaluated. 77 patients excluded either incomplete data or didn't complete both steps within our centers.

ELIGIBILITY:
Inclusion Criteria:

1. patients having stone in the gallbladder and concurrent CBD stone, as determined by MRCP or US.
2. Patients with acute cholecystitis, acute cholangitis, obstructive jaundice, and those with highly suspicious criteria for CBD, stones such as dilated CBD on US examination more than7 mm in diameter without obvious CBD stones, high serum bilirubin level, and or high serum alkaline phosphatase level, were also included in this study.

Exclusion Criteria:

1. Patients with history of hepatobiliary surgery as choledocho-duodenal anastomosis.
2. Patients with previous ERCP attempt.
3. Patients with previous upper abdominal surgery as total or partial gastric resection.
4. Patients with morbid obesity.
5. Patients with uncorrectable coagulopathy.
6. Patients aged below 18 years or above 80 years.
7. Patients within the American Society of Anesthesiology (ASA) class 4 and 5 disease.
8. Patients who refused to give consent or participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
successful stone clearance from the CBD | first year postoperatively
  To ensure that the bile duct was completely clear, a check cholangiogram was conducted.